CLINICAL TRIAL: NCT06749145
Title: Deep Learning Enhanced Detection of Aortic Stenosis - The DETECT-AS-Diagnostic Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Icahn School of Medicine at Mount Sinai (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2000038634; R01AG089981 (NIH)
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Aortic Stenosis
Keywords: aortic stenosis; artificial intelligence
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Intervention (Experimental): The intervention arm will undergo sequential screening for aortic stenosis using portable 1-lead electrocardiograms (ECGs), followed by point-of-care ultrasound (POCUS), if indicated, by artificial intelligence (AI)-based risk algorithms.
  Interventions: Diagnostic Test: Portable 1-lead electrocardiogram; Diagnostic Test: Point-of-care ultrasound; Other: AI-ECG risk algorithm; Other: AI-POCUS
- Control (Sham Comparator): The control arm will undergo a portable 1-lead electrocardiogram (ECG), with 10% randomly assigned to undergo point-of-care ultrasound (POCUS).
  Interventions: Diagnostic Test: Portable 1-lead electrocardiogram; Diagnostic Test: Point-of-care ultrasound

INTERVENTIONS:
Diagnostic Test: Portable 1-lead electrocardiogram — Portable 1-lead electrocardiogram (ECG) performed with the FDA-approved AliveCor KardiaMobile device.
Diagnostic Test: Point-of-care ultrasound — Point-of-care ultrasound performed with the FDA-approved VScan Air device.
Other: AI-ECG risk algorithm — Artificial intelligence (AI) risk algorithm for aortic stenosis using a 1-lead electrocardiogram
  Arms: Intervention
Other: AI-POCUS — Artificial intelligence (AI) risk algorithm for aortic stenosis using cardiac ultrasound plax videos.
  Arms: Intervention

SUMMARY:
The DETECT-AS Diagnostic Study will assess the performance of artificial intelligence (AI) risk predictions to detect aortic stenosis using results from portable electrocardiogram (ECG) and cardiac ultrasound devices.

ELIGIBILITY:
Inclusion Criteria:

* Age 70 years or older
* Attending a routine outpatient primary care clinic at one of the three enrollment sites

Exclusion Criteria:

* Opted out of research studies
* Non-English speaking
* Urgent or emergent visits, defined as a visit for an illness or injury that needs attention quickly or is life-threatening
* Any echocardiogram within 12 months of clinic visit
* Prior history of moderate or severe AS
* Prior history of aortic valve replacement or repair, including transcatheter and surgical AVR with either a bioprosthetic or mechanical valve
* Presence of implantable cardiac devices, including permanent cardiac pacer, implantable cardioverter-defibrillator, or left ventricular assist device
* Prior heart transplant
* History of dementia
* Documented life expectancy of <1 year or current participation in hospice services.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants diagnosed with advanced aortic stenosis (AS) by transthoracic echocardiogram (TTE) | Until 12 months from the baseline visit
  The number of participants diagnosed with advanced AS by TTE at 12 months. Diagnosis of advanced AS is defined as diagnosis of moderate or severe AS as documented in the participant's electronic health record (EHR) at 12 months and adjudication of outcome via review of echocardiographic reports and videos performed by blinded members of the echocardiographic lab at the coordinating center.

CONTACTS AND LOCATIONS:
Overall Officials: Rohan Khera, MD, MS, Principal Investigator — Yale University
Locations (3):
- United States (3):
  - Yale New Haven Health System, New Haven, Connecticut
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - The Methodist Hospital Research Institute, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
A de-identified dataset will be made available following publication of primary results.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code